CLINICAL TRIAL: NCT07011940
Title: Walk With Me (WWM) for Perinatal Grief
Acronym: PeriGrief-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH126788-02; 2R44MH126788-02 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Grief; Post Traumatic Stress Disorder; Suicidal Ideation; Miscarriage; Stillbirth; Infant Death
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation; Abortion, Spontaneous; Stillbirth; Infant Death

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Services as Usual (No Intervention): Services as usual received by referral or identified by the participant
- Along With Me Web-Based Intervention (Experimental): Web-based tool that offers therapeutic support modules with information that leverages cognitive behavioral therapy and mindfulness strategies. The web-based tool includes 10 modules and also includes a list of resources and journaling feature.
  Interventions: Behavioral: Along With Me
- Along With Me Web-Based Intervention Plus Peer Guide Support (Experimental): Web-based tool plus support from a Peer Guide.
  Interventions: Behavioral: Along With Me; Behavioral: Peer Guide

INTERVENTIONS:
Behavioral: Along With Me — Along With Me is a therapeutic app that delivers cognitive behavior therapy and mindfulness-based psychoeducation and skills, grief normalization, and exercises to address perinatal grief and to reduce trauma symptoms related to the experience of perinatal loss. The Along With Me only arm will deliver the app-based intervention only.
  Arms: Along With Me Web-Based Intervention; Along With Me Web-Based Intervention Plus Peer Guide Support
Behavioral: Peer Guide — The peer guide will provide light touch reminders, opportunities to debrief, and resource navigation support, similar to community health navigator interventions provided remotely through insurers.
  Arms: Along With Me Web-Based Intervention Plus Peer Guide Support

SUMMARY:
The goal of this clinical trial is to learn if the Along With Me web-based intervention works to decrease posttraumatic stress symptoms and suicidal ideation among bereaved parents following pregnancy and early infant loss. It will also learn whether peer guides provide additional improvements on these outcomes.

The main questions it aims to answer are:

• Do people who receive Along With Me or Along With Me plus a Peer Guide compared to services as usual have lower posttraumatic stress symptoms and suicidal ideation than those who do not receive the intervention?

Researchers will compare Along With Me and Along With Me plus a Peer Guide to services as usual (referrals made in the hospital setting) to see if Along With Me works to prevent and address posttraumatic stress symptoms and suicidal ideation.

Participants will:

* Receive access to a mobile app with approximately 10 therapeutic modules about how to manage grief and other symptoms.
* Receive check-ins with a Peer Guide (in the Peer Guide condition only)

DETAILED DESCRIPTION:
Our clinical trial is a randomized, three-group controlled trial in which 300 bereaved parents who have experienced pregnancy or early infant loss will be randomly assigned to control (Group 1: treatment as usual, n = 100), Along With Me only (Group 2, n = 100), or the Along With Me Plus Peer Guide (Group 3, n = 100). Participants will be recruited prior to randomization and assigned to condition after consent. Bereaved parents in the treatment arms will receive access to the Along With Me app that provides psychoeducation on grief, and Cognitive Behavioral Therapy (CBT) and Mindfulness skills to manage grief and reduce the risk of posttraumatic stress following pregnancy loss. All participants will complete a baseline assessment that includes self-report of posttraumatic stress symptoms and suicidal ideation, and secondary measures pertaining to mental health symptoms, substance use, coping, grief self-efficacy, and for those in the treatment condition, acceptability and usability for the Along With Me app. Additional assessments will occur at 3 months, 6 months, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Within the first month of pregnancy or early infant loss
* Reside in the United State
* Speak and read either English or Spanish at a 6th grade reading level
* 15 or older

Exclusion Criteria:

* Not pregnant or has not experienced an early infant loss
* Does not reside in the United State
* Does not speak and read either English or Spanish at a 6th grade reading level
* 14 or younger

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline, 3,6,9 months post-baseline
  The PCL-5 is a widely used self-report measure for assessing PTSD symptoms based on Diagnostic and Statistical Manual of Mental Disorders-5 criteria (DSM-5). There are 20 self-report items, and each item is rated on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"). A sum score is computed and can range from 0 to 80, with higher scores indicating greater PTSD symptom severity.
Suicide Cognitions Scale (SCS-R) | Baseline, 3,6,9 months post-baseline
  The SCS-R is a 16-item self-report measure designed to assess suicidogenic cognitions-beliefs and perceptions that increase vulnerability to suicidal behavior. The response option utilizes a 0-4 Likert scale, ranging from 0 (strongly disagree) to 4 (strongly agree). A sum score is computed, resulting in a total score range of 0 to 64. Higher scores indicate stronger endorsement of maladaptive cognitions associated with suicide risk.
Columiba Suicide Severity Rating Scale (C-SSRS) | Baseline, 3, 6, and 9 moths post-baseline
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a 6-item structured set of questions used to assess suicidal ideation (5 items listed from least to most severe) and suicidal behavior (1 item). It is designed to help determine whether suicide-related thoughts/behaviors are present, and if so, their severity and clinical urgency, using standardized definitions and prompts. Response options are on a "yes" and "no" format. Clinically, you use the highest ideation category endorsed (1-5) as the ideation severity indicator and higher scores indicate greater levels of suicidal ideation. The suidial behavior item is a stand alone item indicating presense (=yes) or absence (=no) of any suicidal behavior.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-item scale (GAD-7) | 3, 6, 9 months post-baseline
  The GAD-7 is a 7-item self-report questionnaire designed to screen for and assess the severity of generalized anxiety disorder (GAD). Each item corresponds to one of the core symptoms of GAD as outlined in the DSM-IV. Respondents rate how often they've been bothered by each symptom over the past two weeks using a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total sum score ranges from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.
Patient Health Questionnaire-9 (PHQ-9) | 3,6,9 months post-baseline
  The PHQ-9 is a self-administered tool designed to screen for and measure the severity of depression. It consists of 9 items, each corresponding to one of the DSM-IV criteria for major depressive disorder. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total sum score ranges from 0 to 27, with higher scores indicating greater severity of depression.
Tobacco, Alcohol, Prescription Medication, and Other Substance Use (TAPS) Tool | 3,6,9 months post-baseline
  The TAPS Tool is a brief assessment instrument designed to identify problematic substance use and substance use disorders, consisting of 3-4 items per substance class, evaluating past 3-month usage (=1), problems related to use (=1), and concerns expressed by others (=1). Score for alcohol can range from 0-4, and other substances from 0-3. Scores greater than 1 indicate problematic use, and scores greater than 2 indicate a potential substance use disorder.
Perintal Grief Scale (PGS) | Baseline, 3, 6, and 9 months post-baseline.
  The Perinatal Grief Scale (PGS) is a 33-item brief version was developed to quantify grief reactions following perinatal loss, including losses due to spontaneous abortion, fetal or neonatal death, or ectopic pregnancy. Response options are on a 5-point Likert-type scale (1 = strongly agree, 5 = strongly disagree). All but two items (item 11 and 33) are reveresed scored and three grief subdomain sum scores created: Active Grief (11items), Difficulty Coping (11 items), and Despair (11 items). Subdomain scores can range from 11 to 55 with higher scores indicating higher levels of grief.

CONTACTS AND LOCATIONS:
Overall Officials: David R Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Strategies, Inc., Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be accessible through openICPSR's Search function by topic (e.g., maternal health). Other researchers will be able to see a study description and a link to download data and documentation files. openICPSR provides a DOI number for each data upload such that published study results will be linked to the exact data used and allows depositors to update data files and metadata at any time.
  Survey Data: De-identified individual and aggregate survey data (raw and recoded) will be shared. The de-identification process will remove direct and indirect respondent identifiers. Once data are confirmed final, respondent identifiers will be deleted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Project data and documentation will be uploaded into openICPSR at the time of initial publication, or by the end of the research project period, whichever occurs first. If publication occurs prior to the project's end, researchers will utilize the version update DOI process to maintain data sharing transparency for published study results and supporting data. A complete, deidentified project data set and all supporting documentation will resided on openICPSR as the final data version when the project concludes. Researchers anticipate having project data available in openICPSR for 5 years after the project ends.
Access Criteria: To meet data sharing requirement for our study data and documentation, we have selected the openICPSR repository.